CLINICAL TRIAL: NCT07237789
Title: Impact of Core Stability Training on Function in Patient With Shoulder Impingement Syndrome Among Manual Operated Hand Workers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Salah Eid Ahmed Ali, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SREC.PT.SUE(17)925
Record Dates: First submitted 2025-10-01; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Shoulder Impingement Syndrome
Keywords: Core Stability; Function; Hand Worker; Shoulder Impingement
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Control group will receive traditional physiotherapy
  Interventions: Other: Control
- Experimental (Experimental)
  Interventions: Other: Experimental

INTERVENTIONS:
Other: Experimental — Core stability training will be used for experimental group
  Arms: Experimental
Other: Control — Traditional physiotherapy
  Arms: Control

SUMMARY:
Even at the early stage of employment exposure to mechanical factors such as lifting heavy weights, working with hands at or above shoulder level, and pushing or pulling heavy loads are independent risk factors for new-onset shoulder pain . Shoulder-related problems among workers doing spading are 53.1% and 57.7% among workers brick carrying tasks, these shoulder issues may be the result of repetitive awkward movement (beyond ninety degree raising with abduction position) of the shoulder during these activities .

DETAILED DESCRIPTION:
The highest prevalence of shoulder impingement syndrome is among slaughterhouses as they are exposed to a combination of repetitive shoulder movements and sustained elevated arm .

Several of workplace physical exposures are implicated in the causation and/or increasing shoulder disorders. Occupational exposures including manual handling heavy lifting, pushing, pulling, holding, carrying), working above shoulder height, and repetitive work are the most frequent causes of shoulder disorders specifically the subacromial impingement syndrome.

Shoulder-related problems among workers doing spading are 53.1% and 57.7% among workers brick carrying tasks, these shoulder issues may be the result of repetitive awkward movement (beyond ninety degree raising with abduction position) of the shoulder during these activities.

ELIGIBILITY:
Inclusion Criteria:

manually operated hand workers (males and females), Age from 25-to

-40 years, Shoulder impingement syndrome, and with No previous history of shoulder surgery that may affect their performance.

Exclusion Criteria:

Patient who has a history of shoulder instability, History of shoulder dislocation, Patient who has current symptoms related to the cervical spine, Patient who has a history of acromioclavicular pain, and Low back pain (LBP) will be excluded.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Function | 8 weeks
  DASH-Arabic a self-administered outcome measure will be used to assess disability in patients